CLINICAL TRIAL: NCT06105489
Title: "Tunnel" Flap vs Trapezoidal Flap for Lateral Sinus Lift: A Prospective Randomized Study
Brief Title: "Tunnel" Flap vs Trapezoidal Flap for Lateral Sinus Lift
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Dentistico Associato Sivolella (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20464
Record Dates: First submitted 2023-10-08; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Severe Atrophy of the Edentulous Maxilla
Keywords: Lateral sinus lift; Tunnel technique; Dental Implant; Patient Reported Outcome Measures; Bone Regeneration; Flap Design; Histology; Heterologous bone; Cone Beam Computed Tomography

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two study arms, a test arm and a control arm, for the entire duration of the study.
Masking Description: Health care givers, investigators and outcome assessors cannot be masked to treatment allocation due to the characteristics of the intervention. The statistician will be masked to the treatment allocation during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tunnel flap design (Experimental): Participants will undergo a lateral sinus lift procedure in which a single vertical anterior incision will be made at least 10 mm mesially to the expected outline of the bony window.
  Interventions: Procedure: Lateral Sinus Lift using tunnel flap technique
- Trapezioidal flap design (Active Comparator): Participants will undergo a lateral sinus lift procedure. The incision will be made horizontally on the top of the alveolar ridge, with two additional releasing incisions in the mesial and distal regions.
  Interventions: Procedure: Lateral Sinus Lift using crestal incision flap

INTERVENTIONS:
Procedure: Lateral Sinus Lift using tunnel flap technique — The surgical procedure will involve the following steps:
  * A single vertical anterior incision will be made, at least 10 mm mesially to the expected outline of the bony window.
  * A full-thickness flap will be carefully elevated to expose the lateral wall of the maxillary sinus.
  * A trap door will be created in the lateral wall of the maxillary sinus using either a dedicated piezosurgical insert or a straight handpiece with a 3mm round diamond bur.
  * The door will be removed.
  * The sinus membrane will be gently elevated using various-shaped curettes until it becomes completely detached from the lateral, inferior, and medial walls of the sinus.
  * The maxillary sinus will be filled with a heterologous bone graft with a well-documented efficacy.
  * The flaps will be meticulously sutured.
  Arms: Tunnel flap design
Procedure: Lateral Sinus Lift using crestal incision flap — The surgical procedure will involve the following steps:
  * A horizontal incision is made on the top of the alveolar ridge, along with two additional releasing incisions in the mesial and distal regions.
  * A full-thickness flap will be carefully elevated to expose the lateral wall of the maxillary sinus.
  * A trap door will be created in the lateral wall of the maxillary sinus using either a dedicated piezosurgical insert or a straight handpiece with a 3mm round diamond bur.
  * The door will be removed.
  * The sinus membrane will be gently elevated using various-shaped curettes until it becomes completely detached from the lateral, inferior, and medial walls of the sinus.
  * The maxillary sinus will be filled with a heterologous bone graft with a well-documented efficacy.
  * The flaps will be meticulously sutured.
  Arms: Trapezioidal flap design

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of the lateral sinus lift procedure using the tunnel technique flap in comparison to the traditional lateral sinus lift in partially or totally edentulous patients with loss of teeth in the maxillary premolar or molar areas and severe alveolar atrophy. The primary questions it aims to answer are:

1. Is the tunnel flap technique more suitable for lateral sinus lift than the trapezoidal flap technique in terms of post-operative symptoms?
2. Is the tunnel technique safer and more effective than the trapezoidal flap technique in terms of complication rate and the effectiveness of bone grafting?

Participants will undergo the lateral sinus lift procedure using the tunnel technique, which involves making a vertical anterior incision. Patients will receive follow-up care, including phone contact the day after the procedure to detect any issues, and they will keep a diary during the week after surgery to record visual analog scale (VAS) pain values and analgesics taken. Follow-up surgical visits will be scheduled for suture removal and at 30 days after suture removal. After 6 months, dental implants will be inserted, and prosthetic rehabilitation will take place 6 months later. Implants will be monitored for up to 12 months after prosthetic rehabilitation.

Researchers will compare the outcomes of tunnel flap technique lateral sinus lift with the trapezoidal flap sinus lift.

ELIGIBILITY:
Inclusion Criteria:

* edentulous or partly edentulous patients with a unilateral loss of teeth in the maxillary premolar or molar areas
* severe alveolar atrophy and a residual severe alveolar ridge height up to 3 mm

Exclusion Criteria:

* severe illness
* head and neck radiation therapy
* chemotherapy
* antiresorptive therapy
* uncontrolled diabetes
* uncontrolled periodontal disease
* smoking >10 cigarettes per day
* facial or neck inflammatory or oncologic diseases
* obliteration of sinus ostium and osteomeatal complex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Pain and discomfort on VAS scale at the 4th postoperative day | First week after sinus lift procedure
  Participants will record the subjective post-operative pain/discomfort on a daily VAS score (0 to 10) for the first 7 days, at the same time each day, on a specific form. The VAS is a horizontal ruler 10 cm long with the left end (0 cm) indicating "no pain/discomfort at all" and the right limit (10 cm) indicating "the worst pain imaginable. Patients will be also asked to record the need for analgesics (including type and quantity).

SECONDARY OUTCOMES:
Times for surgical procedure | During sinus lift procedure
  Surgical intervention duration (minutes) recorded from incision to the last suture (T1). Times for sinus mucosa elevation (T2) and for sinus filling (T3) will be measured as well.
Soft tissue healing after sinus lift | 10 days and 40 days after sinus lift procedure
  Soft tissue healing will be evaluated using the scoring reported by Lin SL et al., at two timepoints: at suture removal and at 30 days after suture removal control.
  Assessments of wound healing will include 6 scoring categories, namely erythema, exudate, epithelialization, mucosa color, wound contour, and distortion of mucosa. Each category is scored on a 3-point scale (0, 1, or 2) and a total score from 0 to 3 represents good healing, a score from 4 to 6 represents satisfactory healing, a score from 7 to 9 represents disturbance of healing, and a score from 10 to 12 represents poor healing
Sinus lift related complications | During sinus lift procedure, 1, 10 and 40 days from procedure.
  Possible complications will be evaluated at various timepoints. During the surgical procedure through direct observation (bleeding, sinus membrane perforation, infraorbital nerve injury, perforation of the flap). The day after surgery through a telephone call to the patient (bleeding, flap dehiscence, hematoma, pain). At suture removal control after 10 +/- days after surgery (pain, infections, sinusitis, bone graft displacement, neuropathy, wound dehiscence). At 30 days after suture removal control (pain, infections, sinusitis, bone graft displacement, neuropathy).
Graft healing after a 6 months period | 6 months after implant procedure
  A CBCT of the grafted area finalized to implants insertion planning will be taken after 6 months from the sinus lift. The parameters evaluated will be the final alveolar bone graft height calculated in correspondence of a line passing through the centre of the previous bone window; the presence of the contact between the bone graft and the medial or nasal wall of the sinus cavity; the regular distribution of the graft, intended as the presence of voids or displacements. Moreover a biopsy will be taken during implants insertion by means of a trefine.

OTHER OUTCOMES:
Bone quality | During implant insertion
  Bone quality will be evaluated by means of Lekholm Zarb classification, ranging from D1 for dense cortical bone and D4 for fine trabecular bone.
ISQ and RFA | During implant insertion, 12 months after sinus lift (prosthetic loading), 24 months after sinus lift
  ISQ, ranging from 1 to 100, will be evaluated measuring RFA on two axis (palatal-buccal and mesial-distal) and their mean value will be collected.
Insertion torque | During implant insertion
  Maximum insertion torque will be collected
Peri-implant marginal bone | During implant insertion, 12 months after sinus lift (prosthetic loading), 24 months after sinus lift
  Peri-implant marginal bone variations (mm) will be measured on Periapical radiograph with a standardized technique will be obtained, using methods already described Marginal bone stability (eg Mameno, Tomoaki, et al. "Risk indicators for marginal bone resorption around implants in function for at least 4 years: A retrospective longitudinal study."Journal of periodontology 91.1 (2020): 37-45.)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Sivolella, DDS, PhD, Principal Investigator — Studio Dentistico Associato Sivolella
Locations (1):
- Studio Dentistico Associato Graiff e Sivolella, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyne PJ, James RA. Grafting of the maxillary sinus floor with autogenous marrow and bone. J Oral Surg. 1980 Aug;38(8):613-6. No abstract available. PMID 6993637
- [Background] Stacchi C, Lombardi T, Ottonelli R, Berton F, Perinetti G, Traini T. New bone formation after transcrestal sinus floor elevation was influenced by sinus cavity dimensions: A prospective histologic and histomorphometric study. Clin Oral Implants Res. 2018 May;29(5):465-479. doi: 10.1111/clr.13144. Epub 2018 Mar 23. PMID 29569763
- [Background] Spinato S, Bernardello F, Galindo-Moreno P, Zaffe D. Maxillary sinus augmentation by crestal access: a retrospective study on cavity size and outcome correlation. Clin Oral Implants Res. 2015 Dec;26(12):1375-82. doi: 10.1111/clr.12477. Epub 2014 Sep 5. PMID 25196695
- [Background] Soardi CM, Spinato S, Zaffe D, Wang HL. Atrophic maxillary floor augmentation by mineralized human bone allograft in sinuses of different size: an histologic and histomorphometric analysis. Clin Oral Implants Res. 2011 May;22(5):560-6. doi: 10.1111/j.1600-0501.2010.02034.x. Epub 2010 Dec 9. PMID 21143532
- [Background] Stacchi C, Spinato S, Lombardi T, Bernardello F, Bertoldi C, Zaffe D, Nevins M. Minimally Invasive Management of Implant-Supported Rehabilitation in the Posterior Maxilla, Part II. Surgical Techniques and Decision Tree. Int J Periodontics Restorative Dent. 2020 May/Jun;40(3):e95-e102. doi: 10.11607/prd.4498. PMID 32233185
- [Background] Moy PK, Lundgren S, Holmes RE. Maxillary sinus augmentation: histomorphometric analysis of graft materials for maxillary sinus floor augmentation. J Oral Maxillofac Surg. 1993 Aug;51(8):857-62. doi: 10.1016/s0278-2391(10)80103-x. PMID 8393101
- [Background] Browaeys H, Bouvry P, De Bruyn H. A literature review on biomaterials in sinus augmentation procedures. Clin Implant Dent Relat Res. 2007 Sep;9(3):166-77. doi: 10.1111/j.1708-8208.2007.00050.x. PMID 17716261
- [Background] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Background] Kao SY, Lui MT, Cheng DH, Chen TW. Lateral trap-door window approach with maxillary sinus membrane lifting for dental implant placement in atrophied edentulous alveolar ridge. J Chin Med Assoc. 2015 Feb;78(2):85-8. doi: 10.1016/j.jcma.2014.05.016. Epub 2014 Oct 3. PMID 25287252
- [Background] Silva LD, de Lima VN, Faverani LP, de Mendonca MR, Okamoto R, Pellizzer EP. Maxillary sinus lift surgery-with or without graft material? A systematic review. Int J Oral Maxillofac Surg. 2016 Dec;45(12):1570-1576. doi: 10.1016/j.ijom.2016.09.023. Epub 2016 Oct 17. PMID 27765427
- [Background] Danesh-Sani SA, Engebretson SP, Janal MN. Histomorphometric results of different grafting materials and effect of healing time on bone maturation after sinus floor augmentation: a systematic review and meta-analysis. J Periodontal Res. 2017 Jun;52(3):301-312. doi: 10.1111/jre.12402. Epub 2016 Aug 18. PMID 27534916
- [Background] Stacchi C, Andolsek F, Berton F, Perinetti G, Navarra CO, Di Lenarda R. Intraoperative Complications During Sinus Floor Elevation with Lateral Approach: A Systematic Review. Int J Oral Maxillofac Implants. 2017 May/Jun;32(3):e107-e118. doi: 10.11607/jomi.4884. PMID 28494033
- [Background] Testori T, Weinstein T, Taschieri S, Wallace SS. Risk factors in lateral window sinus elevation surgery. Periodontol 2000. 2019 Oct;81(1):91-123. doi: 10.1111/prd.12286. PMID 31407430
- [Background] Scarano A, Lorusso F, Arcangelo M, D'Arcangelo C, Celletti R, de Oliveira PS. Lateral Sinus Floor Elevation Performed with Trapezoidal and Modified Triangular Flap Designs: A Randomized Pilot Study of Post-Operative Pain Using Thermal Infrared Imaging. Int J Environ Res Public Health. 2018 Jun 16;15(6):1277. doi: 10.3390/ijerph15061277. PMID 29914159
- [Background] Rothstein SS, Paris DA, Zacek MP. Use of hydroxylapatite for the augmentation of deficient alveolar ridges. J Oral Maxillofac Surg. 1984 Apr;42(4):224-30. doi: 10.1016/0278-2391(84)90453-1. PMID 6323657
- [Background] De Stavola L, Tunkel J. Results of vertical bone augmentation with autogenous bone block grafts and the tunnel technique: a clinical prospective study of 10 consecutively treated patients. Int J Periodontics Restorative Dent. 2013 Sep-Oct;33(5):651-9. doi: 10.11607/prd.0932. PMID 23998161
- [Background] Restoy-Lozano A, Dominguez-Mompell JL, Infante-Cossio P, Lara-Chao J, Espin-Galvez F, Lopez-Pizarro V. Reconstruction of mandibular vertical defects for dental implants with autogenous bone block grafts using a tunnel approach: clinical study of 50 cases. Int J Oral Maxillofac Surg. 2015 Nov;44(11):1416-22. doi: 10.1016/j.ijom.2015.05.019. Epub 2015 Jun 23. PMID 26116063
- [Background] Khoury F, Hanser T. Three-Dimensional Vertical Alveolar Ridge Augmentation in the Posterior Maxilla: A 10-year Clinical Study. Int J Oral Maxillofac Implants. 2019 Mar/Apr;34(2):471-480. doi: 10.11607/jomi.6869. PMID 30883623
- [Background] Ponte A, Khoury F. The tunnel technique in bone grafting procedure: A clinical study. Int J Oral Maxxillofac Implants. 2004; 19: 766.
- [Background] Mazzocco C, Buda S, De Paoli S. The tunnel technique: a different approach to block grafting procedures. Int J Periodontics Restorative Dent. 2008 Feb;28(1):45-53. PMID 18351202
- [Background] Restoy A, Pizarro VL, Ordonez V, Lara J, Doussinague BR, Dominguez-Mompell JL. Treatment of the posterior atrophic maxilla using three-dimensional reconstruction technique with sinus lift and a "tunnel" approach. Rev Esp Cir Oral Maxilofac. 2015;37:7-14
- [Background] Lin SL, Wu SL, Tsai CC, Ko SY, Chiang WF, Yang JW. The Use of Solid-Phase Concentrated Growth Factors for Surgical Defects in the Treatment of Dysplastic Lesions of the Oral Mucosa. J Oral Maxillofac Surg. 2016 Dec;74(12):2549-2556. doi: 10.1016/j.joms.2016.06.183. Epub 2016 Jul 1. PMID 27474463